CLINICAL TRIAL: NCT06469996
Title: Effects of Connective Tissue Massage and Self Myofascial Release in Patients With Fibromyalgia
Brief Title: Effects of Connective Tissue Massage in Patients With Fibromyalgia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Firat University (Other)
Responsible Party: Principal Investigator, Songül Bağlan Yentür, Firat University, Firat University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024/08-06
Record Dates: First submitted 2024-06-14; First posted 2024-06-24 (Actual); Last update posted 2024-06-24 (Actual); Status verified 2024-06

CONDITIONS: Fibromyalgia
Keywords: Fibromyalgia; Connective tissue massage; Myofascial release; Foam roller
MeSH Terms: conditions — Fibromyalgia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Connective tissue massage group (Experimental): Connective tissue massage will be applied by an experienced physiotherapist for a total of 12 sessions 2 days a week for 6 weeks. While the patients are in sitting position, starting from the lumbosacral region, the lower thoracic, scapular, interscapular and cervical regions will be included in the treatment respectively.
  Interventions: Other: Connective tissue massage
- Self myofascial relaxation group (Experimental): Self myofascial relaxation will be applied using foam roller. The practice will continue two days a week for 6 weeks. Foam roller exercise is performed in the supine position with knees bent, hands locked behind the neck and foam roller is placed between the shoulder blades.
  Interventions: Other: Self myofascial relaxation

INTERVENTIONS:
Other: Connective tissue massage — Connective Tissue Massage will be applied by an experienced physiotherapist for a total of 12 sessions 2 days a week for 6 weeks. While the patients are in sitting position, starting from the lumbosacral region, the lower thoracic, scapular, interscapular and cervical regions will be included in the treatment respectively.
  Arms: Connective tissue massage group
Other: Self myofascial relaxation — Self myofascial relaxation will be practiced with foam roller in patients with Fibromyalgia.
  Arms: Self myofascial relaxation group

SUMMARY:
Connective tissue massage (CTM), one of the various manual therapy techniques for FMS, produces local mechanical effects on mast cells in the connective tissue with short and long tractions, thereby reducing sympathetic activity and producing vasodilation. The aim of the study was to compare the effectiveness of self myofascial release technique and connective tissue massage in patients with FMS. At least 30 FMS patients will be included in the study. Fibromyalgia Impact Questionnaire, pain, quality of life and sleep quality will be evaluated. CTM will be practiced to study group and foam roller will be practiced to control group.

DETAILED DESCRIPTION:
Fibromyalgia syndrome (FMS) is associated with chronic widespread pain and at least eleven positive tender points out of 18 according to the American College of Rheumatology (ACR) 1990 criteria. It is often associated with symptoms such as decreased physical strength, fatigue, sleep disturbances, gastrointestinal disorders and psychiatric disorders such as depression. Connective tissue massage (CTM), one of the various manual therapy techniques for FMS, produces local mechanical effects on mast cells in the connective tissue with short and long tractions, thereby reducing sympathetic activity and producing vasodilation. In the last two decades, massage applications using tools of various densities, materials, shapes and sizes (such as Foam Roller (FR), roller massagers, sticks or balls) and actively self-administered by individuals have rapidly gained popularity. The aim of the study was to compare the effectiveness of self myofascial release technique and connective tissue massage in patients with FMS. At least 30 FMS patients will be included in the study. Fibromyalgia Impact Questionnaire, pain, quality of life and sleep quality will be evaluated. CTM will be practiced to study group and foam roller will be practiced to control group. Treatments will be applied for 6 weeks, 2 days a week for a total of 12 sessions.

ELIGIBILITY:
Inclusion Criteria:

* Being a woman
* Being diagnosed with FMS,
* Being between the ages of 18-65 and volunteering.

Exclusion Criteria:

* Neurological, infectious, endocrine and other inflammatory rheumatic diseases, severe psychological disorders, any condition that prevents exercise (advanced cardiac respiratory or orthopedic problems),
* Malignancy
* Being pregnant

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-06-20 (Estimated); Primary Completion 2024-08-20 (Estimated); Study Completion 2024-08-30 (Estimated)

PRIMARY OUTCOMES:
disability | 2 minutes
  Fibromyalgia Impact Questionnaire is a scale consisting of 10 questions to assess the health status and physical functionality of an individual diagnosed with FM.

SECONDARY OUTCOMES:
pain assesment | 1 minute
  Pain will be evaluated with Visual Analog Scale. Patients will be asked to rate the severity of pain between 0-10.
Quality of life assesment | 2 minutes
  Quality of life will be assessed with the Health Assessment Questionnaire (HRA). The HRA is one of the first disability questionnaires used in adults with arthritis. The highest scores of each subgroup are summed and the result is divided by eight to obtain the participant's SDQ score.

CONTACTS AND LOCATIONS:
Locations (1):
- Songul, Elâzığ, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No